CLINICAL TRIAL: NCT00746174
Title: Insulin Resistance and Intramyocellular Lipid Content in Glucose Intolerant Subjects Receiving Rosiglitazone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Lidia S. Szczepaniak, PhD., University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSK CRT49653/250
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Insulin Sensitivity
Keywords: insulin sensitivity; magnetic resonance spectroscopy (MRS); lipotoxicity; lipid oxidation; thiazolidinediones; intracellular; triglyceride; content
MeSH Terms: conditions — Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosiglitazone (Active Comparator): Subjects in this arm will be randomly assigned to treatment with Rosiglitazone 4mg daily. After 4 weeks, we will assess changes in glucose levels and liver enzymes. The dose will then be increased to Rosiglitazone 8mg daily (if indicated). The patients will be reevaluated every 4 weeks, and at the end of 16 weeks, the participants will all be admitted to the research center at UTSW to measure changes in the following: 1) insulin sensitivity; 2) lipid content of heart, liver, & skeletal muscle; and 3) lipid oxidation using respiratory gas exchange. The patients will then switch to the alternative therapy for 16 additional weeks before the studies are repeated.
  Interventions: Drug: Rosiglitazone
- Placebo (Placebo Comparator): Subjects in this arm will be randomly assigned to treatment with placebo. After 4 weeks, we will assess changes in glucose levels and liver enzymes. The patients will be reevaluated every 4 weeks, and at the end of 16 weeks, the participants will all be admitted to the research center at UTSW to measure changes in the following: 1) insulin sensitivity; 2) lipid content of heart, liver, & skeletal muscle; and 3) lipid oxidation using respiratory gas exchange. The patients will then switch to the alternative therapy for 16 additional weeks before the studies are repeated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — Rosiglitazone 8mg PO daily for 16 weeks
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Placebo — Placebo 1 tablet PO daily for 16 weeks
  Arms: Placebo

SUMMARY:
This study will include subjects with an abnormal glucose tolerance test. Using a crossover design, we will evaluate the insulin sensitivity and intracellular lipid content of the heart, liver and skeletal muscle of subjects before and after therapy with Rosiglitazone and placebo. We hypothesize that Rosiglitazone will improve insulin sensitivity in association with reduced muscle lipid content that may arise either from increased lipid oxidation or enhanced storage of fat in adipose tissue.

DETAILED DESCRIPTION:
This protocol is a crossover study that will include subjects with an abnormal glucose tolerance test. Participants will be treated in a community-based practice setting and will receive detailed instruction on diet and glucose self-monitoring. The patients will be randomly assigned to treatment with 4 mg daily of Rosiglitazone or placebo. They will return to the clinic after 4 weeks to monitor changes in glucose levels, HbA1c and liver enzymes. The drug dose will be increased as indicated to 8 mg daily and the patients will be reevaluated every 4 weeks. The participants will all be admitted to the General Clinical Research Center at UT-Southwestern Medical Center at the end of 16 weeks to measure changes in the following primary endpoints: 1) insulin sensitivity, 2) lipid content of heart, liver, and skeletal muscle, 3) lipid oxidation. Additional noninvasive HMRS measurements will be made to quantify the muscle lipid content and respiratory gas exchange will be used to assess lipid oxidation. Following the GCRC admission, patients will switch to the alternative therapy for 16 additional weeks before the studies are repeated. We expect Rosiglitazone to improve insulin sensitivity in association with reduced muscle lipid content that may arise either from increased lipid oxidation or enhanced storage of fat in adipose tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65
* Fasting plasma glucose < 126 mg/dL or plasma glucose > 140 mg/dL and <200 mg/dL two hours after a challenge with 75 gm of glucose

Exclusion Criteria:

* Taking drugs known or suspected to affect intermediary metabolism (e.g. thyroid supplements, oral glucocorticoids, anabolic steroids or androgens, antidepressants, anorexic drugs, xanthine derivatives, sympathomimetics, beta-agonists)
* Taking any other investigational drugs within 30 days of starting the study
* Alcohol consumption more than 7 drinks per week
* Recreational drugs or IV drug abuse
* Acute or chronic liver diseases (SGOT >42 U/L, SGPT >48 U/L, GGT >45 U/L)
* Chronic renal insufficiency (serum creatinine >1.5 mg/dL)
* Uncontrolled hypertension (systolic/diastolic blood pressure >160/95mmHg)
* Anemia (hematocrit <35%)
* Congestive heart failure
* Metallic prostheses precluding the use of magnetic resonance imaging
* Premenopausal women without definitive measures to prevent pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 16 weeks

SECONDARY OUTCOMES:
Intracellular lipid content in myocardium, liver and skeletal muscle | 16 weeks
Lipid oxidation | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lidia S Szczepaniak, PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States